CLINICAL TRIAL: NCT05976438
Title: Investigating the Relevance of Skin Sodium and Salt Sensitivity of Blood Pressure in Determining the Response to Anti-Hypertensive Drugs (INTREPID)
Brief Title: Skin Sodium and Salt Sensitivity of Blood Pressure
Acronym: INTREPID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Prof, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A096461
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
Keywords: Skin Sodium; Salt Sensitivity; Blood Pressure; Heart Disease; Cardiovascular
MeSH Terms: conditions — Hypertension; Heart Diseases | interventions — Amlodipine; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open label arm 1 (Other): Participants will be randomised to AB sequence of drugs A: 1 to 2 weeks of Amlodipine 5mg followed by 6 to 7 weeks of Amlodipine 10mg B: Approximately 8 weeks of 25mg Chlortalidone
  Interventions: Drug: Amlodipine; Drug: Chlortalidone
- Open label arm 2 (Other): Participants will be randomised to BA sequence of drugs B: Approximately 8 weeks of 25mg Chlortalidone A: 1 to 2 weeks of Amlodipine 5mg followed by 6 to 7 weeks of Amlodipine 10mg
  Interventions: Drug: Amlodipine; Drug: Chlortalidone

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5mg and Amlodipine 10mg will be one of the study drugs the patients will receive.
Drug: Chlortalidone — Chlortalidone 25mg will be one of the study drugs the patients will receive.

SUMMARY:
Eating too much salt raises blood pressure and the risk of having a heart attack or stroke. The investigators do not fully understand why salt raises blood pressure, but storage of sodium in the body, particularly in the skin, may be important. For this reason, the investigators wish to study the link between skin sodium, blood pressure and cardiovascular risk in patients with high blood pressure, of different ethnicities, using techniques such as skin biopsy and magnetic resonance imaging (MRI). The results will provide detailed information on skin sodium storage and help us better understand the effects of blood pressure medications on these mechanisms. Ultimately, the investigators aim to develop personalized treatment guidelines for clinical use.

DETAILED DESCRIPTION:
The physiological basis of salt sensitivity of blood pressure (SSBP) is poorly understood, and determining which patients have SSBP is not straightforward. Furthermore, determining salt sensitivity requires direct intervention tracking changes in blood pressure after salt challenge or depletion over several days. This makes identifying salt-sensitive individuals impractical in a clinical setting, hindering its application. It is crucial that the investigators elucidate the underlying mechanisms of salt-sensitivity, and through this understanding develop a biomarker of SSBP for clinical use.

From a review of recent studies it appears that in the short-term, accumulation of skin sodium during high salt intake attenuates the blood pressure response, while in the long-term, high skin sodium levels indicate a tendency for SSBP, hypertension and elevated cardiovascular risk. The reasons for this are not clear and merit further investigation. By refining methods for quantification of skin sodium and expanding its use in hypertension research, the clinicians can improve patient assessment, treatment prescription, and disease monitoring.

Using skin biopsy and sodium MRI provides a unique opportunity to study skin sodium handling and SSBP during antihypertensive treatment, and can provide insights into why hypertensives and certain ethnic groups have a higher incidence of SSBP. Sodium MRI may also help increase our understanding of the mechanisms by which diuretics work, both systemically and in the kidney and provide a way to identify salt-sensitive individuals for targeted clinical intervention.

Hypotheses:

1. Skin sodium decreases with salt-dependent (diuretic) treatments but not salt-independent (calcium channel blocker) treatments.
2. Diuretic-induced reductions in skin sodium correlate with reductions in blood pressure.
3. Skin sodium is higher in populations traditionally known to be more salt sensitive, such hypertensive patients of black ethnicity.

Patients will be enrolled on to a randomised, open-label, two-treatment two-period crossover treatment. The hypertensive medication used in this study are Amlodipine 5 or 10mg and Chlortalidone 25mg.

The duration for individual participants will be approximately 16 weeks. Participants will have a total of 7 visits including screening/enrolment (visit 1) and baseline visit (visit 2).

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent to participate
2. Aged 18 or above
3. Be hypertensive defined as:

   1. Currently untreated with an ABPM day time average blood pressure or average home blood pressure of ≥135 mmHg (systolic) or ≥85 mmHg (diastolic)

      OR
   2. Patients who are taking antihypertensive drugs at sub therapeutic doses or in ineffective combinations, and who are felt likely to be controllable on a study drug and willing and able to be washed out, at the discretion of the CI/PI, can enter the study if they meet the above criteria.

Exclusion Criteria:

1. Uncontrolled blood pressure ≥ 180/110mmHg
2. Known or suspected secondary hypertension
3. Pregnant or breastfeeding women
4. Significant sensitivity or contraindications to any of the study medications
5. Participants taking lithium or are regularly consuming non-steroidal anti-inflammatory drugs at variable doses
6. Requirement to take any of the study drugs continuously e.g. ACEi and heart failure
7. Any clinically significant hepatic impairment
8. Any clinically significant kidney impairment
9. Concurrent participation in another clinical trial or study using systemic vasoactive medications or medications known to interact with the study drugs
10. Patients who are deemed unsuitable by the investigator on clinical grounds e.g. an abnormal heart rhythm due to Atrial Fibrillation (AF)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of Skin sodium | Approximately 8 weeks after receiving each treatment up to week 16 which will be the study completion week
  This is planned for all participants
Concentration of Skin Potassium | Approximately 8 weeks after receiving each treatment up to week 16 which will be the study completion week
  This is planned for all participants
Systolic blood pressure | All study visits - every 4 weeks up to week 16 which will be the study completion week
  This is planned for all participants

SECONDARY OUTCOMES:
MRI skin sodium concentration | Approximately 8 weeks after receiving each treatment up to week 16 which will be the study completion week
  This is planned for all participants
Concentration of Skin glycosaminoglycans | Approximately 8 weeks after receiving each treatment up to week 16 which will be the study completion week
  This is planned for all participants
Diastolic blood pressure | All study visits - every 4 weeks up to week 16 which will be the study completion week
  This is planned for all participants
Body weight | Body weight measurement will be performed at baseline only.
  This is planned for all participants

OTHER OUTCOMES:
Sodium MRI of kidney | Approximately 8 weeks after receiving each treatment up to week 16 which will be the study completion week
  This is planned for patients who consent to sodium imaging of kidney

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - St Thomas' Hospital, London